CLINICAL TRIAL: NCT00079547
Title: The Safety and Efficacy of Low and High Carbohydrate Diets
Brief Title: The Safety and Effectiveness of Low and High Carbohydrate Diets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT001103-01 (NIH); R01AT001103-01 (NIH)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
Keywords: Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Caloric Restriction; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Low-calorie diet
  Interventions: Behavioral: Low-calorie diet
- 2 (Experimental): Low-carbohydrate diet
  Interventions: Behavioral: low-carbohydrate diet

INTERVENTIONS:
Behavioral: Low-calorie diet — low-calorie diet
  Arms: 1
Behavioral: low-carbohydrate diet — low-carbohydrate diet
  Arms: 2

SUMMARY:
This study will compare the safety and the effectiveness of a low carbohydrate diet (Atkins diet) with a high carbohydrate diet (conventional USDA diet).

DETAILED DESCRIPTION:
Despite the considerable mass appeal of popular diet books, such diet approaches lack data to support their efficacy and safety. Despite its widespread use for more than 30 years, the Atkins diet has never been evaluated in a large, randomized, controlled trial. This study will assess the short-term and long-term clinical effects of a low-carbohydrate diet and a high-carbohydrate diet in overweight and obese men and women.

Participants in this study will be randomly assigned to the Atkins diet (low-carbohydrate, unlimited fat and protein) or a conventional USDA diet (high-carbohydrate, low-fat). The study will evaluate the effects of each dietary approach on changes in: 1) weight and body composition; 2) metabolic and organ function; and 3) exercise tolerance. Each participant will be enrolled in the study for 2 years.

ELIGIBILITY:
Inclusion Criteria

* Body mass index between 30 and 40
* Live and work within 1 hour of the study site
* Stable psychological status

Exclusion criteria

* History of heart disease, heart attack, or stroke
* Blood pressure >140/90 mmHg
* Abnormal cholesterol levels
* Significant psychiatric illness
* Any medication that affects weight or metabolic rate
* Presence or history of a chronic disease that is known to affect appetite, food intake, or metabolism (i.e., diabetes, thyroid disease, or cancer)
* Currently using antidepressants, steroids, tobacco, or illegal drugs
* Pregnant, breastfeeding, or planning pregnancy
* 10 lb change in weight within 6 months of study entry
* History of malignant arrhythmias or cerebrovascular, renal, or hepatic disease
* History of protein wasting diseases or gout
* Severe arthritis
* Osteoporosis
* Certain types of hormone replacement therapy
* Currently following a vegetarian diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2003-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
weight change | 2 years

SECONDARY OUTCOMES:
change in lipids | 2 years
blood pressure change | 2 years
Ketones | 2 years
Endothelial Function | 2
change in exercise endurance | 2 years
change in renal function | 2 years
change in bone density | 2 years
change in body composition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — University of Pennsylvania; Holly Wyatt, MD, Principal Investigator — University of Colorado, Denver; James Hill, PhD, Principal Investigator — University of Colorado, Denver; Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] de las Fuentes L, Waggoner AD, Mohammed BS, Stein RI, Miller BV 3rd, Foster GD, Wyatt HR, Klein S, Davila-Roman VG. Effect of moderate diet-induced weight loss and weight regain on cardiovascular structure and function. J Am Coll Cardiol. 2009 Dec 15;54(25):2376-81. doi: 10.1016/j.jacc.2009.07.054. PMID 20082927